CLINICAL TRIAL: NCT06473103
Title: Investigation of Standard Excision Surgical Margins Using Two Photon Fluorescence Microscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Rochester Dermatologic Surgery (Other)
Responsible Party: Principal Investigator, Michael Giacomelli, Associate Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00009521
Record Dates: First submitted 2024-06-07; First posted 2024-06-25 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- TPFM imaging of surgical margins (Experimental): Excised tissue will be imaged with TPFM to determine the distance from tumor to nearest inked margin.
  Interventions: Device: Two photon fluorescence microscopy imaging

INTERVENTIONS:
Device: Two photon fluorescence microscopy imaging — Excised tissues will be imaged with two photon fluorescence microscopy prior to submission for histological processing.

SUMMARY:
The goal of this clinical trial is to compare the use of two photon fluorescence microscopy for detecting residual basal cell carcinoma during standard local excision.

DETAILED DESCRIPTION:
This study is an study of skin cancer that will evaluate the feasibility of two photon fluorescence microscopy (TPFM) to evaluate surgical margins followed by standard of care permanent sections for final margin confirmation. To protect patients, following TPFM imaging, patients will receive standard of care evaluation on permanent sections, thus all patients will receive standard of care confirmation following experimental imaging. Individual excisions from consenting patients will be selected, fluorescently labeled and the distance to inked margins measured with TPFM. Following imaging, specimens will be submitted for paraffin processing as per normal procedure and the resulting slides scanned. The distance to the inked margin will be measured on the permanent sections and compared to TPFM to determine accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing treatment for basal cell carcinoma without Mohs surgery at the performance site
* Able to read and understand consent form

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Quantitative agreement between clear margin distance on TPFM and conventional paraffin embedded histology | Upon receipt of postoperative pathology slides, typically 2-4 weeks post surgery
  The distance from the furthest extent of the tumor to the nearest surgical margin will be measured on both TPFM and conventional paraffin histology and the numerical difference calculated.

SECONDARY OUTCOMES:
Overall agreement on margin status | Upon receipt of postoperative pathology slides, typically 2-4 weeks post surgery
  The status of margins (positive/negative) will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Michael Giacomelli, Principal Investigator — University of Rochester
Locations (1):
- Rochester Dermatologic Surgery, Victor, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ching-Roa VD, Huang CZ, Ibrahim SF, Smoller BR, Giacomelli MG. Real-time Analysis of Skin Biopsy Specimens With 2-Photon Fluorescence Microscopy. JAMA Dermatol. 2022 Oct 1;158(10):1175-1182. doi: 10.1001/jamadermatol.2022.3628. PMID 36069886